CLINICAL TRIAL: NCT02398708
Title: Comparison of the Fecal Microbiome, Peripheral Inflammatory Markers, and Symptoms in Individuals Discordant for GVHD After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Comparison of Gut Microbiota, Inflammation and Symptoms Following Allogeneic HSCT
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400992; UF-BMT-cGVHD-101 (Other: University of Florida Protocol ID); ID00023244 (Other Grant/Funding Number: American Cancer Society); OCR14208 (Other: OnCore)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Graft vs Host Disease; Graft Versus Host Disease; Hematopoietic Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation
Keywords: Hematopoietic Stem Cell Transplantation; Graft versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and stool specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Graft-Versus-Host Disease: This group will have questionnaires, clinical data, a blood sample and a stool sample collected to be compared with the other group.
  Interventions: Other: Questionnaires; Other: Blood Sample; Other: Stool Sample; Other: Clinical data
- No Chronic Graft-Versus-Host Disease: This group will have questionnaires, clinical data, a blood sample and a stool sample collected to be compared with the other group.
  Interventions: Other: Questionnaires; Other: Blood Sample; Other: Stool Sample; Other: Clinical data

INTERVENTIONS:
Other: Questionnaires — Both groups will have questionnaires collected and compared.
Other: Blood Sample — Both groups will have a blood sample collected and compared.
Other: Stool Sample — Both groups will have a stool sample collected and compared.
Other: Clinical data — Both groups will have clinical data collected and compared.

SUMMARY:
The purpose of this study is to examine the gut bacteria, levels of peripheral blood inflammation markers, and symptoms in patients with and without chronic graft-versus-host disease (cGVHD) following allogeneic hematopoietic stem cell transplant (allo-HSCT). The hypothesis is that individuals with cGVHD will have lower levels of microbial diversity, higher levels of inflammatory metabolites in stool and peripheral measures, and higher levels of symptoms than individuals without cGVHD.

DETAILED DESCRIPTION:
This study will recruit 40 (20 with cGVHD and 20 without cGVHD) adults from the Bone Marrow Transplant Program at University of Florida Health Shands Cancer Hospital. After signing informed consent, participants will fill out questionnaires and have a blood sample collected from a vein in the arm. Participants will be given a stool collection kit with instruction and will return the sample via the mail. Data will be collected and securely stored in a system used by the cancer center for research. Descriptive statistics will be used to report individual, clinical factors, and symptoms.

Knowledge gained from this study will provide preliminary data for future longitudinal studies to examine biological pathways for the development, severity and/or duration of cGVHD and symptom outcomes in individuals following allo-HSCT impacting quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Adults (> 18 years of age) within 3 months to 3 years of receiving allogeneic hematopoietic stem cell transplant (allo-HSCT) diagnosed with cGVHD;
* Group 2: Adults (> 18 years of age) within 3 months to 3 years of receiving allo-HSCT without a diagnosis of cGVHD; and
* All participants must be able and willing to complete paper and pencil questionnaires, provide a blood and stool sample, and be able to give informed consent.

Exclusion Criteria:

* Diagnosed with a significant secondary inflammatory disease such as multiple sclerosis, Crohn's disease, rheumatoid arthritis or secondary cancer;
* History of a major psychological disorder requiring psychotropic medications or initiation of antidepressants within 30 days of enrollment;
* Incarcerated or pregnant; or
* Any other condition that in the opinion of the principal investigator (PI) may compromise study participation will not be eligible for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 allo-Hematopoietic Stem Cell Transplantation (HSCT) recipients with chronic graft-versus-host disease (cGVHD) and 20 allo-Hematopoietic Stem Cell Transplantation (HSCT) recipients without chronic graft-versus-host disease (cGVHD)
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Plasma levels of inflammatory markers (cytokines and CRP) of individuals post allogeneic HSCT | Day 1
  Cytokines will be analyzed using a multiplex assay by Millipore Company. Compared to the traditional enzyme-linked immunosorbant assays (ELISA), the multiplex is comparable and more sensitive to lower concentration levels of cytokines than the ELISA. One laser identifies a specific bead and another laser identifies the reported antibody associated with the bead-bound cytokine. One hundred beads for each of the 17 cytokines in every sample are assayed and a mean cytokine binding for the sample is determined. The manufacturer reports that the assay accurately measures cytokine values in a range of 1-2500pg/ml. Serum CRP will be measured using the ALPCO's (American Laboratory Products Company) high-sensitivity CRP assay which uses latex particle enhanced immunoturbidimetry for quantitative CRP determination.
Diversity and levels of fecal microbes of individuals post allogeneic HSCT | Day 1
  Fecal microbial DNA will be extracted from between 50-200 mg of fecal material. The 16S ribosomal gene (V4 region) of each sample will be amplified using a barcoding system to allow multiplexing with the Illumina MiSeq system. We will use UNIFRAC algorithm to evaluate the null hypothesis that the structure of the microbial community is insensitive to cGVHD and symptoms of cGVHD. Differences in taxa are implicated by our high throughput sequencing methods will be confirmed by other techniques including culturing (where appropriate) and qPCR with taxa-specific primers.
Behavioral responses (symptoms) of individuals post allogeneic HSCT | Day 1

SECONDARY OUTCOMES:
Health Promoting Lifestyle Profile II (HPLPII) | Day 1
  The Health Promoting Lifestyle Profile II (HPLPII) will be used to identify lifestyle choices that may affect relationships and differences between groups. HPLPII measures health promoting behaviors across several dimensions with subscales of health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations and stress management. This is a 52-item summated behavior rating scale using a 4-point response format to measure the frequency of self-reported health-promoting behaviors. It is a well validated toll and takes approximately 10 minutes to complete.
Perceived Stress Scale (PSS) | Day 1
  The Perceived Stress Scale (PSS) will be used to measure individual's level of perceived stress which may affect levels of inflammation. This is a short 10 question form rating individuals ability to tolerate change and unpredictable situations. This is the most widely used measure of individual's perceived stress and is well validated. It takes approximately 5 minutes to complete.
Brief Pain Inventory (BPI) | Day 1
  Pain will be assessed using the Brief Pain Inventory (BPI). The BPI was created to evaluate two dimensions of pain: 1) the severity and 2) the interference. This tool is well validated with Cronbach's alpha .80-.87 pain severity and .89-.92 for interference.22 The BPI consists of a body diagram to indicate location of pain and a general question asking if pain is present. Four items assess pain intensity or severity and seven item s assess pain interference. Both use an eleven point scale ranging from 0 (no pain or interference) to 10 (worst pain or interference). This instrument takes approximate five minutes to complete.
Hospital Anxiety and Depression Scale (HADS) | Day 1
  Depressive symptoms will be assessed using the subscale for depression from the Hospital Anxiety and Depression Scale (HADS). 23This instrument is used to assess the presence and severity of anxiety and depressive symptoms over a seven day period. The depression subscale is comprised of seven items using a four point scale ranging from 0 (least severe) to 3 (most severe). Cronbach's alpha has been found to be high (.82-.90) for the HADS depression subscale.
Brief Fatigue Inventory (BFI) | Day 1
  Fatigue will be assessed using the Brief Fatigue Inventory (BFI). The BFI is a nine item, eleven point scale that assesses physical, affective, cognitive and social domains in a two dimensions, fatigue intensity and interference. Severity scores are as follows: 1) mild (1-3), 2) moderate (4-6) and 3) severe (7-10). This tool is well establish and validated. The Cronbach's alpha ranged from .95-.96 for individual items and an internal consistency of .96 overall. The questionnaire takes approximately five minutes to complete and a global score can be ascertained by averaging the total score.
Lee Symptom Bother Scale | Day 1
  The Lee Symptom Bother Scale is a multi-symptom scale that measures the severity of symptoms as described as how much a symptom bothers the patient. 25There are seven domains assessed: 1) skin, 2) eye, 3) mouth, 4) lung function, 5) nutrition, 6) psychosocial status, and 7) energy. All areas are rated using a 5 point Likert type scale where 0 indicates "Not at all" and 4 indicates "Extremely" bothered. A summary score is created by taking the mean of all items and linearly transforming that value to a 0-100 scale. The Chronbach's α is between .79 and .90. The test-retest reliability for all subscales is .74-.93 except psychosocial is .55 and lung is .28. The scale has good convergent validity.
Memorial Symptom Assessment Scale (MSAS-SF) | Day 1
  To comprehensively explore symptoms, the Memorial Symptom Assessment Scale (MSAS-SF) will be used to measure multiple dimensions (frequency, severity, and distress) of 32 common cancer symptoms. The Cronbach alpha for the MSAS-SF subscales ranged from .76-.86 and the test-retest correlation coefficients ranged from .86-.94 at one day and one week respectively. The total time to complete this form is approximately 10 minutes. This form allows for patients to identify and quantify "other" symptoms.
Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) | Day 1
  Health related quality of life (HRQOL) will be measured using the Functional Assessment of Cancer Therapy- Bone Marrow Transplantation (FACT-BMT). This is a well validated HRQOL measure. This is a 27-item questionnaire asking questions across four domains: physical well-being, social well-being, emotional well-being and functional well-being. This measure takes about 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lynch Kelly, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Hospital, Gainesville, Florida, United States